CLINICAL TRIAL: NCT06361550
Title: Effectiveness of a Nutritional Intervention in Improving the Mediterranean Diet in Older Adults
Brief Title: Nutritional Status Assessment and Dietary Recommendations Program (VENREDI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Ayuntamiento de Salamanca (Unknown)
Responsible Party: Principal Investigator, Fausto Jose Barbero-Iglesias, Principal investigation, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AYTO_SALAMANCA_001
Record Dates: First submitted 2024-04-03; First posted 2024-04-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Adherence to the Mediterranean Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Practical seminar, carried out in a market, on how to properly carry out the shopping cart. Afterwards, the participants will prepare a menu, consisting of three courses (starter, main and dessert). Finally, the tasting of the different preparations will take place.
  Interventions: Other: VENREDI group
- Control (Active Comparator): Group educational talk, lasting 2 hours, aimed at correct compliance with the Mediterranean Diet according to current recommendations.
  Interventions: Other: Health education

INTERVENTIONS:
Other: VENREDI group — Practical seminars aimed at improving the Mediterranean diet, guided by researchers.
  Arms: Intervention group
Other: Health education — Health education on Mediterranean diet
  Arms: Control

SUMMARY:
Introduction: The Mediterranean diet has been related to beneficial effects in the prevention of cardiovascular diseases and other chronic pathologies related to diet, including some types of cancer. Specifically in the elderly population, it has been observed that the Mediterranean diet is inversely associated with all causes of mortality and that the greater the adherence to this type of diet, the lower the mortality in elderly adults.

Objective: To evaluate the effect of a multifactorial intervention (seminar on shopping basket and food labeling, workshop on healthy cooking and subsequent tasting of the prepared products) in improving adherence to the Mediterranean diet in older adults.

Methodology: Randomized controlled clinical trial with two parallel groups: an intervention group (IG) and a control group (CG). The study population will be adults over 60 years of age, retired or pre-retired. A sample size of 200 participants has been estimated, 100 in each group to detect a difference of 0.83 points or more in the MEDAS questionnaire.

All participants will receive an educational talk on healthy nutrition, with an estimated duration of 2 hours. The GI, in addition to this educational workshop, will receive a practical seminar on how to properly carry out the shopping cart. This will take place both in a market and later in a supermarket in Salamanca. In addition, a workshop will be held where participants will prepare a menu consisting of three dishes (starter, main and dessert) and will later taste them.

An initial and post-intervention evaluation will be carried out after 3 months so that both groups can study the change variables related to Adherence to the Mediterranean Diet [Mediterranean Diet Adherence Questionnaire (MEDAS)], physical activity [Short physical performance battery (SPPB)], sleep quality (ATENAS questionnaire) and assessment of cognitive function (MOCA questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years old, retired or in early retirement
* Participate in the program "Research in active aging with preventive physiotherapy - PReGe"
* Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Present any pathology that prevents carrying out the workshops appropriately.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to the Mediterranean Diet | Baseline, 3 months
  Mediterranean Diet Adherence Questionnaire (MEDAS). Minimum [Worse] 0 - Maximum [Better] 14

SECONDARY OUTCOMES:
Physical activity | Baseline, 3 months
  Short Physical Performance Battery. Minimum [Worse] 0 - Maximum [Better] 12
Sleep Quality | Baseline, 3 months
  Atenas questionnaire. Minimum [Better] 0 - Maximum [Worse] 24
Cognitive function | Baseline, 3 months
  MOCA questionnaire. Minimum [Worse] 0 - Maximum [Better] 30

CONTACTS AND LOCATIONS:
Locations (1):
- Rosario Alonso Domínguez, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No